CLINICAL TRIAL: NCT03583346
Title: A Phase Ib, Single-center, Double-blind, Randomized, Placebo-controlled, Parallel-group, Multiple Ascending Dose Study to Assess Safety, Tolerability, Immunogenicity, Pharmacokinetics, and Pharmacodynamics of Subcutaneous Injections of M6495 (Anti-ADAMTS-5 Nanobody) in Participants With Symptomatic Knee Osteoarthritis
Brief Title: Multiple Ascending Doses (MAD) of Anti-A Disintegrin and Metalloproteinase With Thrombospondin Motifs-5 (Anti-ADAMTS-5) Nanobody in Participants With Knee Osteoarthritis (OA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS200572_0003; 2018-000797-29 (EudraCT Number)
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Osteoarthritis, Knee
Keywords: M6495; Anti-ADAMTS-5 Nanobody; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M6495 (Experimental)
  Interventions: Drug: M6495
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: M6495 — Participants will receive escalated dose of M6495 bi-weekly on Day 1, 15 and 29 in cohort 1 to 3 and weekly on Day 1, 8, 15, 22, 29 and 36 in cohort 4.
  Arms: M6495
Drug: Placebo — Participants will receive placebo matched to M6495 bi-weekly on Day 1, 15 and 29 in cohort 1 to 3 and weekly on Day 1, 8, 15, 22, 29 and 36 in cohort 4.
  Arms: Placebo

SUMMARY:
The study will be conducted in participants with symptomatic knee OA to explore the safety, tolerability, immunogenicity, pharmacokinetics (PK), and pharmacodynamics (PD) of MAD of M6495.

ELIGIBILITY:
Inclusion Criteria:

* Kellgren Lawrence (KL) radiological Grade of 2 to 4 in the target knee
* Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscore of greater than or equal to (>=) 40 out of 100 in the target knee at screening
* Primary or post-traumatic femorotibial OA according to American College of Rheumatology clinical and radiographic criteria
* Have completed at least 4 days of the participant 7-day diary in the period from Day -8 to Day 1
* Can give signed informed consent
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* History of arthroscopy or intra-articular administration of corticosteroids or hyaluronic acid into the target knee within 6 months before screening
* Intention of having major knee surgeries or total knee replacement during the time frame of this study in either knee
* Secondary OA in target knee joint because of joint dysplasia, aseptic osteonecrosis, acromegaly, Paget disease, Stickler syndrome, hemochromatosis, gout, chondrocalcinosis, or calcium pyrophosphate deposition disease
* Any known active systemic infection, including infection that might compromise the immune system such as human immunodeficiency virus, or hepatitis B or C
* History of myocardial infarction or cerebrovascular event within 6 months prior to screening, or current active angina pectoris, symptomatic heart failure, seizures, untreated hypertension, gastrointestinal bleeding, or any other significant medical condition in the Investigator's opinion
* History of cancer, except adequately treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ/cervical intraepithelial neoplasia of the uterine cervix, unless considered cured >= 5 years
* Other protocol defined exclusion criteria could apply

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Occurrences of Treatment-emergent Adverse Events (TEAEs), Treatment-related AEs and Serious AEs (SAEs) | Day 1 up to Day 106
Number of Participants With Clinically Significant Change From Baseline in Vital Signs, Laboratory Parameters and 12-lead Electrocardiogram (ECG) Findings | Day 1 up to Day 106
  Number of participants with clinically significant change from baseline will be reported.
Occurrences of Injection Site Reactions | Day 1 up to Day 43

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of M6495 | Day 1 up to Day 106
Dose Normalized Maximum Serum Concentration (Cmax/Dose) of M6495 | Day 1 up to Day 106
Accumulation Ratio for Cmax (Racc [Cmax]) of M6495 | Day 1, 15 and 29
  Following Racc parameters will be measured:
  * Racc15 (Cmax): Cmax at Day 15/Cmax at Day 1
  * Racc29 (Cmax): Cmax at Day 29/Cmax at Day 1
Immunogenicity of M6495 as Assessed by Antidrug Antibodies (ADA) Assays | Day 1 up to Day 106

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- DanTrials ApS, Copenhagen NV, Denmark